CLINICAL TRIAL: NCT06503679
Title: A Phase 1, Single-center, Open-label, Fixed-sequence, Crossover Study to Evaluate the Effect of LY4100511 (DC-853) on the Single-dose Pharmacokinetics of Midazolam, Repaglinide, Digoxin, and Rosuvastatin in Healthy Participants
Brief Title: A Drug-drug Interaction Study Evaluating the Perpetrator Potential of LY4100511 (DC-853) on Midazolam, Repaglinide, Digoxin, Rosuvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27110; J5C-MC-FOAF, DC-853104 (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company)
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: LY4100511; DC-853
MeSH Terms: interventions — Midazolam; repaglinide; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY4100511 Dose 1 + Midazolam + Repaglinide (Cohort 1) (Experimental): Participants will receive an oral dose 1 of LY4100511 and single dose of midazolam and repaglinide.
  Interventions: Drug: LY4100511 (DC-853) Dose 1; Drug: Midazolam; Drug: Repaglinide
- LY4100511 Dose 2 + Midazolam + Repaglinide (Cohort 2) (Experimental): Participants will receive up to an oral dose 2 of LY4100511 and single dose of midazolam and repaglinide. Dosing will not proceed until a satisfactory review of the safety and tolerability data from lower dose level is performed.
  Interventions: Drug: LY4100511 (DC-853) Dose 2; Drug: Midazolam; Drug: Repaglinide
- LY4100511 Dose 3 + Digoxin and Rosuvastatin (Cohort 3) (Experimental): Participants will recive an oral dose 3 of LY4100511 and single dose of digoxin and rosuvastatin.
  Interventions: Drug: LY4100511 (DC-853) Dose 3; Drug: Digoxin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: LY4100511 (DC-853) Dose 1 — Administered orally
  Arms: LY4100511 Dose 1 + Midazolam + Repaglinide (Cohort 1)
Drug: LY4100511 (DC-853) Dose 2 — Administered orally
  Arms: LY4100511 Dose 2 + Midazolam + Repaglinide (Cohort 2)
Drug: LY4100511 (DC-853) Dose 3 — Administered orally
  Arms: LY4100511 Dose 3 + Digoxin and Rosuvastatin (Cohort 3)
Drug: Midazolam — Administered orally
  Arms: LY4100511 Dose 1 + Midazolam + Repaglinide (Cohort 1); LY4100511 Dose 2 + Midazolam + Repaglinide (Cohort 2)
Drug: Repaglinide — Administered orally
  Arms: LY4100511 Dose 1 + Midazolam + Repaglinide (Cohort 1); LY4100511 Dose 2 + Midazolam + Repaglinide (Cohort 2)
Drug: Digoxin — Administered orally
  Arms: LY4100511 Dose 3 + Digoxin and Rosuvastatin (Cohort 3)
Drug: Rosuvastatin — Administered orally
  Arms: LY4100511 Dose 3 + Digoxin and Rosuvastatin (Cohort 3)

SUMMARY:
The main purpose of this study is to assess the safety and tolerability and pharmacokinetics of LY4100511 (DC-853) when administered alone or in the presence of cytochrome P450 substrates in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Females must be of childbearing potential
* Males must agree to use contraception
* Have body mass index (BMI) between 18.0 and 32.0 kilogram/square meter (kg/m²), inclusive, and a body weight of greater than or equal to 50 kg.
* In good health, as determined by no clinically significant findings from medical history, 12-lead ECG and vital signs measurements, and clincial laboratory evaluations (congentical nonhemolytic hyperbilirubinemia) at screening and check-in, and from the physical examination at check-in as assessed by the investigator.

Exclusion Criteria:

* Have a 12-lead ECG abnormality that, in the opinion of the investigator,

  * increases the risks associated with participating in the study
  * may confound ECG data analysis
  * a QTCF >450 msec for males, or >470 msec for females

    * short PR interval <120 msec or PR interval >220 msec
    * second or third degree atrioventricular block
    * intraventricular conduction delay with QRS >120 msec
    * complete right bundle branch block
    * left bundle branch block, or
    * Wolff Parkinson-White syndrome.
* Have had current or recent acute infection
* Show evidence of active or latent tuberculosis (TB)
* Had any surgical procedures within 12 weeks prior to screening or any planned surgical procedure scheduled to occur during the study.
* Have a history or presence of multiple or severe allergies, or an anaphylactic reaction to prescription or non prescription drugs.
* Are immunocompromised
* Presence of active suicidal ideation or positive suicide behavior using baseline/screening version of the C-SSRS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC [0-∞]) of Midazolam, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
Pharmacokinetics (PK): Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC [0-∞]) of 1-Hydroxymidazolam, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
Pharmacokinetics (PK): Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC [0-∞]) of Repaglinide, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
Pharmacokinetics (PK): Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC [0-∞]) of Digoxin, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
PK: Area Under the Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC[0-tlast]) of Midazolam, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
PK: Area Under the Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC[0-tlast]) of 1-Hydroxymidazolam, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
PK: Area Under the Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC[0-tlast]) of Repaglinide,in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
PK: Area Under the Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC[0-tlast]) of Digoxin, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
PK: Maximum Observed Concentration (Cmax) of Midazolam, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
PK: Maximum Observed Concentration (Cmax) of 1-Hydroxymidazolam, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
PK: Maximum Observed Concentration (Cmax) of Repaglinide, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose
PK: Maximum Observed Concentration (Cmax) of Digoxin, in the absence or presence of steady-state LY4100511 | Day 1 and Day 9: Predose, Up to 48 Hours Post Dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No